CLINICAL TRIAL: NCT00469768
Title: A Double-blind, Randomized, Placebo-controlled Safety and Pharmacokinetic Study in Healthy HIV-negative Women to Assess the Delivery of Dapivirine From Matrix and Reservoir Intravaginal Rings Each Containing 25 mg of Dapivirine
Brief Title: A Pharmacokinetic Study of Dapivirine Vaginal Rings in Belgium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Zeda Rosenberg ScD, International Partnership for Microbicides
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 018
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: dapivirine matrix intravaginal ring
- B (Experimental)
  Interventions: Drug: dapivirine reservoir intravaginal ring
- C (Placebo Comparator)
  Interventions: Other: placebo intravaginal ring

INTERVENTIONS:
Drug: dapivirine reservoir intravaginal ring — a silicone elastomer reservoir ring containing 25mg of dapivirine
  Arms: B
Drug: dapivirine matrix intravaginal ring — a silicone elastomer matrix intravaginal ring containing 25mg of dapivirine
  Arms: A
Other: placebo intravaginal ring — a silicone elastomer intravaginal ring containing no dapivirine
  Arms: C

SUMMARY:
IPM 018 is a double-blind, randomized, placebo-controlled study conducted at one site in Belgium among 24 healthy, HIV-negative women to evaluate dapivirine release for 28 days from matrix and reservoir intravaginal rings, each containing 25 mg of dapivirine, and to assess safety and tolerability compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 35 years of age
* Willing and able to give written informed consent
* Available for all visits and consent to follow all procedures scheduled for the study
* Healthy and HIV-negative as determined by a HIV-1 ELISA test at time of enrollment;
* Willing to abstain from sexual activity for the duration of the study
* Willing to use oral contraceptives to avoid menstruation while taking part in this study or on long-acting progestins for 6 months prior to enrollment
* Upon pelvic / speculum examination at enrollment, the cervix and vagina appear normal
* Willing to refrain from use of vaginal products or objects for the duration of the study.

Exclusion Criteria:

* History of alcoholism, drug abuse, psychosis, antagonistic personality, poor motivation, or other emotional or intellectual problems that are likely to invalidate the informed consent process or adversely impact compliance with protocol requirements;
* History of sensitivity / allergy to latex, dapivirine or to the constituents of the vaginal ring (i.e. silicone elastomer)
* Currently pregnant or breast-feeding, or within three months of last pregnancy outcome
* Currently or within one month of participating in any other clinical research study
* History or diagnosis of and / or treatment for a sexually transmitted disease within the last three months
* History of genital tract surgery within the last month
* Current diagnosis of sexually transmitted infections (Gonorrhea, Chlamydia and Trichomonas)
* Current vulvar or vaginal symptoms / abnormalities that could influence the study results
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding or urethral obstruction within the last three months;
* Smoking more than 10 cigarettes per day

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Annalene Nel, Study Director — International Partnership for Microbicides (IPM)
Locations (1):
- Drug Research Unit Ghent (D.R.U.G.), Ghent, Belgium